CLINICAL TRIAL: NCT06853223
Title: A Randomized Trial of CCR5 Inhibition as a Complement to Lung Transplant Induction Immunosuppression
Brief Title: This Study is Assessing the Safety and Efficacy of Immune Inhibition as a Treatment to Prevent Primary Graft Dysfunction
Acronym: MARAVIROC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-43392
Record Dates: First submitted 2025-02-14; First posted 2025-02-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Primary Graft Dysfunction; Lung Transplantation; Acute Lung Injury(ALI); Natural Killer Cell Mediated Immunity
MeSH Terms: conditions — Primary Graft Dysfunction; Acute Lung Injury | interventions — Maraviroc

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled phase 2 study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Maraviroc (Experimental): This arm is the Maraviroc drug which will be administered to patients.
  Interventions: Drug: Maraviroc
- Placebo (Placebo Comparator): This arm is the placebo drug which will be matched in appearance and taste to the Maraviroc and is available in PO and liquid (PFT) formulations.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maraviroc — Product will be administered for 300 mg immediately preceding the lung transplant surgery and then will be administered every 12 hours. There will be 7 total doses. The first 3 will be 300 mg doses and the remaining 4 will be 150 mg doses. Maraviroc will be given oral (PO) or by feeding tube (PFT) in crushed format depending on the route availability.
  Arms: Maraviroc
Drug: Placebo — Placebo in 300 and 150 mg formulations Product will be administered every 12 hours for 3 days. The placebo will be matched in appearance and taste to the Maraviroc and is available in PO and liquid (PFT) formulations.
  Arms: Placebo

SUMMARY:
Lung transplant recipient survival lags other solid organ recipients, with the main early cause of death being primary graft dysfunction (PGD). PGD occurs in up to 1/3 of all recipients, is driven by the body's innate immune response, and has no known medical therapies for treatment or prevention. Investigators have recently shown that Natural Killer (NK) cells, a key innate immune cell, are critical in causing PGD. Importantly, the investigators found that Maraviroc, an FDA-approved drug that works to inhibit these immune cells, prevented lung injury in mouse models of PGD.

The goal of this clinical trial is to learn if Maraviroc works to treat PGD in Lung Transplant patients who are above the age of 18 and have a PGD risk score greater than 50%. The objectives the study hopes to address are:

To address the safety and tolerability of Maraviroc. To test a strategy for PGD enrichment in a lung transplant population. To measure the efficacy and biological efficacy of using Maraviroc. To study the biochemical, physiologic, and molecular effects of the drug on the body.

This will be a double blind study where patients will either get the Maraviroc drug or a placebo. Researchers will then compare the two groups to address the above objectives.

Participants will:

Take drug Maraviroc or a placebo every 12 hours for 3 days post surgery. Follow up will occur during the entire length of stay at UCSF, about 16 days, with a single 12 month follow up once released.

DETAILED DESCRIPTION:
This trial seeks to pilot processes to optimize for a multi-center clinical trial of CCR5 inhibition before transplant. Investigators will measure success in enriching a lung transplant population for PGD and will investigate the feasibility of recruitment for a pilot trial of CCR5 inhibition. Investigators will also assess the safety and tolerability of CCR5 inhibition in lung transplant recipients. Investigators will measure key adverse events and assess for drug-drug interactions. In addition, investigators will measure Maraviroc drug levels in plasma and bronchoalveolar lavage to determine dosing efficacy. Increasingly, there is awareness that subphenotypes of diseases exist and can be leveraged for targeted therapies. Therefore, the investigators also seek to develop standard assays for future subphenotyping efforts in a larger multicenter clinical trial. To do this, the investigators will measure donor and recipient biologic endpoints. These include bronchoalveolar lavage NK cells after transplant as a surrogate marker for biologic efficacy.

A complete physical examination will be performed by either the investigator or a sub investigator who is a physician at Baseline/Screening Visit 1. Qualified staff (MD, NP, RN, and PA) may complete the abbreviated physical exams at all other visits. New abnormal physical exam findings must be documented and will be followed by a physician or other qualified staff at the next scheduled visit. The experimental product, Maraviroc, will be administered in 300mg and 150mg formulations. Product will be administered for 300 mg in the PACU and then will receive doses every 12 hours with 2 additional 300 mg doses and the remaining will be 150 mg doses for a total of 7 doses over 3 days. Maraviroc will be given oral (PO) or by feeding tube (PFT) in crushed format depending on the route availability. Placebo will be administered in a reflective capacity and in similar dosage. Patients will be in the study for up to 28 days, all of which will be during their hospital stay, leading up to and following their lung transplant operation. A final subject follow up will occur 12 months later. When approximately 50% of patients have completed the study through Visit 6, an interim analysis for safety will be conducted by an independent data monitoring committee.

The association between the maraviroc treatment group and placebo control group and severe PGD (primary endpoint) or continuous secondary endpoints (such as immune populations) will be tested using logistic or linear regression, respectively. For study's secondary analysis of maximum PGD grade, investigators will use cumulative linked models assessing PGD as an ordinal variable. All models will be adjusted for variables that may introduce clinical heterogeneity (age, sex, ethnicity, transplant type, transplant indication) and are not established PGD risk factors or used in the randomization tool. Each endpoint/experimental aim will work from a fixed cohort of 30 participants randomized to CCR5 inhibition (maraviroc group, n = 15) or placebo control (placebo group, n = 15). Investigators will use an enrichment tool to target an incidence of PGD of 50% in our study population. Conservatively, it is expected that approximately 75% of the consented cohort will not meet randomization criteria. Thus, there will be 90 consented participants with <50% risk for PGD to be used as clinical comparators (Low risk PGD group). For the investigator's primary outcome, it is expected that 80% power will detect an estimated effect size of 0.39 with a two-tailed alpha of 0.051. This equates to a power to resolve a difference in 9.5% in severe PGD between treatment and control groups. These effect sizes provide ample power for the primary outcomes of interest based on previously reported data within the field.

Complete blood counts (hemoglobin, hematocrit, red blood cell count, white blood cell count, white blood cell differential, and platelet count) are measured per routine clinical care. Investigators will record the baseline CBC obtained near the time of lung transplant waitlisting as well as CBCs performed on post-operative days (POD) 0-3, POD 7, POD14, and POD30. Serum sodium, potassium, chloride, bicarbonate, random glucose, BUN, creatinine, aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), alkaline phosphatase, total bilirubin, direct bilirubin, tacrolimus trough, and posaconazole levels are also collected as part of routine clinical care. These data points from the time nearest to lung transplant waitlisting as a baseline as well as chemistries performed on POD 0-3, POD 7, POD14, and POD30 will be recorded. Blood for determination of serum concentrations of maraviroc will be collected pre-dose as well as at 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72, 84, and 96 hours after the start of dosing. Investigators will collect vials of blood for plasma banking pre-dose and on POD 1 and POD 3 and store/ process it in a lung transplant biorepository according to established protocols.

Investigators will perform a lavage of the donor lung during back table OR preparation with 20 mL of saline. Bronchoscopy for routine graft assessment occurs at the bedside on POD 0 through 3. During the POD 1 and POD 3 bronchoscopies, we will perform lavage in the right middle lobe or lingula with 20 mL of saline. Specimens will be collected in a sterile 50 mL falcon tube. The tube will be labeled, packed in ice and transferred to our laboratory for processing. Investigators plan to perform BAL cell immunophenotyping with spectral flow cytometry, BAL supernatant cytokine measurements, and will bank cell pellets in qiazol for future RNA sequencing. The data will be entered into a validated UCSF RedCap database. The PI will be responsible for data processing, in accordance with procedural documentation. Database lock will occur once quality assurance procedures have been completed. All procedures for the handling and analysis of data will be conducted using good computing practices meeting FDA guidelines for the handling and analysis of data for clinical trials. After data have been entered into the study database, a system of computerized data validation checks will be implemented and applied to the database on a regular basis. The study database will be updated in accordance with the resolved queries. All changes to the study database will be documented.

This is a single center pilot study. As such, there is no appointed "Medical Monitor." Rather, the study PI (Dr. Calabrese) and co-Investigator (Dr. Hays) should be contacted directly at these numbers to report medical concerns or questions regarding safety. Subjects may be discontinued from study treatment at any time if the subject, the investigator, or the Sponsor feels that it is not in the subject's best interest to continue. This may be due to a subject withdrawal of consent, the emergence of adverse events that in the opinion of the investigator would be in the best interest of the subject to discontinue study treatment, or if a protocol violation requires discontinuation of study treatment. If a subject is withdrawn from treatment due to an adverse event, the subject will be followed and treated by the Investigator until the abnormal parameter or symptom has resolved or stabilized. All subjects who discontinue study treatment will be evaluated in the hospital for an early discontinuation visit as soon as possible and then should be encouraged to complete all remaining scheduled visits and procedures. All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice. Reasonable attempts will be made by the investigator to provide a reason for subject withdrawals.

The study will have an independent Data and Safety Monitoring Board (DSMB) that will advise and periodically monitor participant safety and evaluate the progress of the study. The DSMB will review all changes to the study plan and will review procedures for maintaining data confidentiality, data integrity, and data analyses. The DSMB has not been selected yet for this study, but participants will be recruited from inside UCSF and outside of the institution. The board will have a range of specialties and backgrounds to account for the complexity of the patient population. The DSMB will meet quarterly to review study progress, data quality and participant safety. Safety reports will be sent 2 weeks before each meeting to afford statistical overview and review beforehand. De-identified but unmasked data will be provided to the DSMB statistician for data processing and analysis. Raw data identifying individual participants will not be available to the DSMB. After the conclusion of the study, the DSMB will confer with the study team to provide individual participants' health providers with pertinent information from the trial. The study team will discuss results with each randomized trial participant after all data has been analyzed but before publication of results. The data and safety monitoring reports will contain both masked and unmasked data. Reports will be generated with the help of the DSMB statistician. A report template has been created and will be available for the DSMB to review. Unmasking will be provided at written request from the DSMB statistician to the Investigational Pharmacy Service. Patient data will remain deidentified throughout the data analysis process. The reports will include information on the study status, participant enrollment status, participant descriptive information, and data on adverse events and serious adverse events by organ system. While some summary tables will show unmasked treatments, data will be presented in a blinded manner during open DSMB meetings. All data and discussion inside DSMB will be confidential. The responsibilities of the DSMB and individual voting members are outlined in the IRB. The DSMB will meet quarterly through the end of the patient phase of the study and then twice annually. The DSMB will propose additional analyses and discuss the rationale for continuation of the study or stopping early for safety. At the end of each DSMB, the group will vote on whether to continue the study and make recommendations on proposed protocol changes. The DSMB will also review data integrity at each meeting and review manuscripts of trial results as requested by the trial team.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at the time of lung transplant waitlisting.
2. Listed for a bilateral lung transplantation.
3. Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
4. PGD risk score > 50% at the time of donor organ offer
5. Planned induction with basiliximab, mycophenolatge, and prednisone and routine maintenance immunosuppression of tacrolimus, mycophenolate and prednisone.

Exclusion Criteria:

1. Recipient scheduled to receive alternate induction regimen that is cell depleting such as anti-thymocyte globulin or alemtuzumab.
2. Active chronic pulmonary infection in the recipient that are considered relative contraindications to lung transplantation such as Burkholderia or Mycobacterium abscessus.
3. Recipients receiving HIV, HCV or HBV positive donor organs. Only documented infections are considered exclusion criteria. Recipients receiving increased risk organs will not be excluded.
4. Recipient listed for concurrent heart or other solid organ transplantation.
5. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-07 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-08-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe Primary Graft Dysfunction | 3 days

SECONDARY OUTCOMES:
Post-operative outcomes associated with PGD | 3 months
  Will compare the time to extubation from mechanical ventilation (time in minutes)
Other measures of Primary Graft Dysfunction | 3 days
  Maximum PGD grade on post-operative day 0-3.
Biologic markers of efficacy. | 12 months
  Proportion and absolute count of bronchoalveolar lavage NK cells
Mortality within first year | 12 months
  If death occurs within the first year of transplant.
Measures of allograft function | 12 months
  Investigators will track incidents of chest imaging findings.
Other measures of Primary Graft Dysfunction. | 3 days
  Lowest PaO2/FiO2 (P/F ratio) on PD 0-3.
Other measures of Primary Graft Dysfunction | 12 months
  PaO2/FiO2 (P/F ratio) as a continuous outcome variable.
Other measures of Primary Graft Dysfunction | 12 months
  Incidence of post-operative extracorporeal membranous oxygenation (ECMO) need.
3. Biologic markers of efficacy. | 12 months
  Proportion and absolute count of bronchoalveolar lavage CCR5+ lymphocytes
Biological markers efficacy | 12 months
  Proportion and absolute count of BAL CCR5+ NK cells
Measures of allograft function | 12 months
  Investigators will track FEV1 (in absolute Liters)
Measures of allograft function | 12 months
  Investigators will track Maximum FVC (absolute liters)
Post-operative outcomes associated with PGD | 3 months
  Post-operative lengths of stay (time in days) for the intensive care unit.
Post-operative outcomes associated with PGD | 3 months
  Post-operative lengths of stay (time in days) for the patient's general hospital stay to those of non PGD patients

OTHER OUTCOMES:
Maraviroc PK evaluations | 4 days
  We will measure maraviroc levels in plasma (ng/mL) at pre-dose and then every 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Calabrese, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No